CLINICAL TRIAL: NCT05789342
Title: A Four-part, Single-center, Open-label, Phase I Clinical Study to Evaluate the Drug-drug Interactions (DDIs) Between GP681 and Rosuvastatin/Digoxin/Itraconazole/Oseltamivir in Chinese Healthy Volunteers
Brief Title: A Study to Evaluate the Drug-drug Interactions (DDIs) of GP681 With Rosuvastatin, Digoxin, Itraconazole, Oseltamivir in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP681-202202
Record Dates: First submitted 2023-02-21; First posted 2023-03-29 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Rosuvastatin Calcium; Digoxin; Itraconazole; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The DDI of GP681 and Rosuvastatin Calcium Tablets (Experimental): Subjects will receive a single dose of Rosuvastatin Calcium 10 mg on Day 1, then take a single doses of 40mg GP681, 10mg Rosuvastatin Calcium on Day 8.
  Interventions: Drug: GP681; Drug: Rosuvastatin
- The DDI of GP681 and Digoxin Tablets (Experimental): Subjects will receive a single dose of Digoxin 0.25 mg on Day 1, then take a single doses of 40mg GP681, 0.25mg Digoxin on Day 15.
  Interventions: Drug: GP681; Drug: Digoxin
- The DDI of GP681 and Itraconazole Capsules (Experimental): Subjects will receive a single dose of GP681 20mg on Day 1, then take Itraconazole 200 mg twice-daily on Day 22 and 200 mg once-daily on Day 23 through Day 36, and took a single dose of GP681 20 mg on Day 26.
  Interventions: Drug: GP681; Drug: Itraconazole
- The DDI of GP681 and Oseltamivir Capsules (Experimental): Subjects will receive all three treatments in a crossover fashion according to the randomized sequence. The treatments were as follows: single oral administration of GP681 at 40 mg on day 1 in the fasted state; single oral administration of oseltamivir at 75 mg on day 1 and day 5in the fasted state, followed by repeated twice-daily administration of oseltamivir at 75 mg until day 5 after each meal; co-administration of GP681 at 40 mg and oseltamivir at 75 mg simultaneously on day 1 in the fasted state, followed by repeated twice-daily administration of oseltamivir at 75 mg until day5 after each meal. There was an at least 21-day washout interval between each treatment.
  Interventions: Drug: GP681; Drug: Oseltamivir

INTERVENTIONS:
Drug: GP681 — GP681, tablet, oral
Drug: Rosuvastatin — Rosuvastatin, tablet, oral
  Arms: The DDI of GP681 and Rosuvastatin Calcium Tablets
Drug: Digoxin — Digoxin, tablet, oral
  Arms: The DDI of GP681 and Digoxin Tablets
Drug: Itraconazole — Itraconazole, capsule, oral
  Arms: The DDI of GP681 and Itraconazole Capsules
Drug: Oseltamivir — Oseltamivir, capsule, oral
  Arms: The DDI of GP681 and Oseltamivir Capsules

SUMMARY:
This study is a four-part, single-center, Open label phase I clinical study to characterize the DDIs potential of GP681 With Rosuvastatin, Digoxin, Itraconazole or Oseltamivir in Chinese healthy volunteers. This study also aims to evaluate the safety and tolerability of GP681 in the presence of Rosuvastatin, Digoxin, Itraconazole, or Oseltamivir.

DETAILED DESCRIPTION:
GP681 is a potent polymerase acidic (PA) protein endonuclease inhibitor. This study will be run in four parts to characterize the DDIs potential of GP681 with the expected concomitant drugs (Rosuvastatin, Digoxin, Itraconazole, Oseltamivir) in Healthy Subjects. Each part of this study consists of a screening period (Day -14 to Day -1), a baseline period (Day -1), a treatment period, and a follow-up telephone call for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females between the ages of 18 and 55 years, inclusive;
2. Body weight ≥50.0 kg for males, ≥45kg for females, and body mass index (BMI) between19-26 kg/m^2(inclusive);
3. Normal physical examination, vital signs, 12-lead ECG, Chest X-ray images (anteroposterior) and clinical laboratory values, or any abnormality that is non-clinically significant;
4. Men must agree to use protocol-specified contraception and also to not donate sperm throughout the study and for at least 3 months after the final dose of study drug
5. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions.

Exclusion Criteria:

1. History of allergic conditions or allergic diseases, or a history of allergic reactions attributed to GP681 or any of the ingredients of its formulation or similar drugs. Those who cannot follow a uniform diet for special dietary requirements.
2. Subjects with swallowing difficulties, or have diseases such as hemorrhoids, perianal diseases with regular/bleeding in the stool, habitual constipation or diarrhea, irritable bowel syndrome and inflammatory bowel diseases, affecting drug absorption, distribution, metabolism, excretion or the efficacy and safety of the drug.
3. History of gastrointestinal ulcer or bleeding; Or history of any clinically significant diseases or diseases which may affect the result of this study, such as gastrointestinal, circulatory, respiratory, endocrine, neurological, urinary, hematological, immunological, psychiatric and metabolic diseases;
4. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsade de pointes ventricular tachycardia, ventricular tachycardia, prolonged QT syndrome, or symptoms of prolonged QT syndrome and family history;
5. Patients who have undergone surgery within 6 months before the screening period, or who have undergone major surgery within 28 days, or whose surgical incision is not completely healed; Major surgery includes, but is not limited to, any surgery with a significant risk of bleeding, prolonged general anesthesia, or an open biopsy or significant traumatic injury;
6. Pregnant or lactating female subjects, female subjects with childbearing potential and positive pregnancy test at baseline.
7. History of receiving a live vaccine within 1 month prior to the screening, or is expected to receive a live vaccine during the study.
8. Any positive test result of hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody;
9. Received any drugs that inhibit or induce the CYP450 enzyme (i.e., inducers-barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors- SSRI-antidepressant, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines) 30 days prior to screening period;
10. Received any drugs (including Chinese herbal medicine, vitamins and supplements) within 14 days prior to dosing, or participation in another clinical trial within 3 months before dosing.
11. Those who have lost blood or donated up to 200 mL within 3 months before dosing, or those who plan to donate blood within 1 month after the end of this study;
12. Smoking more than 5 cigarettes per day within 3 months prior to screening，or who cannot stop using any tobacco products during the study period;
13. Average weekly intake of alcohol is more than 21 units alcohol (1 units ≈ 360 mL beer, or 45 mL spirits with 40% content, or 150 mL wine) within the 3 months prior to dosing, or a positive ethanol breath test at screening;
14. Substance abuse or use of soft drugs (e.g., marijuana) or use of hard drugs (e.g., cocaine, amphetamines, phenylcyclohexidine, etc.); Or screening for positive urine drug abuse (drug) tests;
15. Habitual or excessive consumption (more than 8 cups, 1cup=250mL) of grapefruit juice, tea, coffee and/or caffeinated beverages;
16. Subjects who are intolerant to venipuncture or have a history of fainting blood or acupuncture
17. Inability to take normal hospital diet;
18. Subjects with poor compliance, or not suitable for this study as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Part one: Peak plasma concentration (Cmax) of Rosuvastatin | Day 1 to Day 4, and Day 8 to Day 11
Part one: Area under the plasma concentration versus time curve (AUC) of Rosuvastatin | Day 1 to Day 4, and Day 8 to Day 11
Part two: Peak plasma concentration (Cmax) of Digoxin | Day 1 to Day8, and Day 15 to Day 22
Part two: Area under the plasma concentration versus time curve (AUC) of Digoxin | Day 1 to Day 8, and Day 15 to Day 22
Part three: Peak plasma concentration (Cmax) of GP681 | Day 1 to Day12, and Day26 to Day 37
Part three: Area under the plasma concentration versus time curve (AUC) of GP681 | Day 1 to Day 12, and Day26 to Day 37
Part Four: Peak plasma concentration (Cmax) of GP681 | 264 hours after GP681 administration
Part Four: Area under the plasma concentration versus time curve (AUC) of GP681 | 264 hours after GP681 administration
Part Four: Peak plasma concentration (Cmax) of Oseltamivir | 12 hours after Oseltamivir administration
Part Four: Area under the plasma concentration versus time curve (AUC) of Oseltamivir | 12 hours after Oseltamivir administration

CONTACTS AND LOCATIONS:
Overall Officials: Jintong Li, Principal Investigator — China-Japan Friendship Hospital; Gang Cui, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han M, Cui G, Zhao Y, Zuo X, Wang X, Zhang X, Mi N, Jin J, Xiao C, Wang J, Wu W, Li Y, Li J. Evaluation of drug-drug interaction between Suraxavir Marboxil (GP681) and itraconazole, and assessment of the impact of gene polymorphism. Front Pharmacol. 2025 Apr 11;15:1505557. doi: 10.3389/fphar.2024.1505557. eCollection 2024. PMID 40291342